CLINICAL TRIAL: NCT03002662
Title: Cecal Intubation Time in Colonoscopy: Prospective Clinical Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ebubekir Gündeş, Gastroenterogical Surgery, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Other Study IDs: 2016.5/8-19
Record Dates: First submitted 2016-12-18; First posted 2016-12-26 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-05

CONDITIONS: Endoscopy; Colonoscopy
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (4):
- BMI <18.5 underweight (Group 1): BMI was calculated as weight in kilograms divided by the square of height in meters. BMI <18.5 underweight (Group 1)
  Interventions: Other: colonoscopy
- BMİ: 18.5 - 24.9 normal weight (Group 2): BMI was calculated as weight in kilograms divided by the square of height in meters. BMİ: 18.5 - 24.9 normal weight (Group 2)
  Interventions: Other: colonoscopy
- BMİ: 25- 29.9 overweight (Group 3): BMI was calculated as weight in kilograms divided by the square of height in meters. BMİ: 25- 29.9 overweight (Group 3)
  Interventions: Other: colonoscopy
- BMİ>30 obese (Group 4): BMI was calculated as weight in kilograms divided by the square of height in meters. BMİ>30 obese (Group 4)
  Interventions: Other: colonoscopy

INTERVENTIONS:
Other: colonoscopy

SUMMARY:
During colonoscopy, body mass index, waist circumference and waist / hip ratio is the relationship between the cecal intubation difficulty aims to define.

ELIGIBILITY:
Inclusion Criteria:

1. Above 18

Exclusion Criteria:

1. Bad bowel preparation
2. Failure of cecum intubation
3. Inflammatory bowel disease
4. Colectomy story

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are cases of distant referral to the gastroenterology surgeon's polyclinic and indications for colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-09-01 (Estimated); Study Completion 2017-09-15 (Estimated)

PRIMARY OUTCOMES:
Body mass index (kg/m2) | 12/01/2016- 05/01/2017
waist circumference (centimeter) | 12/01/2016- 05/01/2017
waist / hip ratio | 12/01/2016- 05/01/2017

CONTACTS AND LOCATIONS:
Locations (1):
- Eagle Run High Special Education and Research Hospital, Istanbul, Turkey (Türkiye)